CLINICAL TRIAL: NCT00679952
Title: Randomised Prospective Study of Clinical Outcomes After Closed Suction Drainage and Natural Drainage of the Pancreatic Duct in Pancreaticojejunostomy After Pancreatoduodenectomy
Brief Title: Closed Suction Drainage and Natural Drainage of the Pancreatic Duct in Pancreaticojejunostomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-0612-018-191
Record Dates: First submitted 2008-05-15; First posted 2008-05-19 (Estimated); Results first posted 2011-05-09 (Estimated); Last update posted 2014-05-19 (Estimated); Status verified 2014-05

CONDITIONS: Pancreatic Fistula
Keywords: Pancreatic fistula; Pancreatic duct stent; Closed suction drainage
MeSH Terms: conditions — Pancreatic Fistula | interventions — Pancreaticojejunostomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): closed suction drainage group (CD group)
  Interventions: Procedure: closed suction drainage of pancreatic duct
- 2 (Active Comparator): natural drainage group (ND group)
  Interventions: Procedure: natural drainage of pancreatic duct

INTERVENTIONS:
Procedure: closed suction drainage of pancreatic duct — A Fr 5-8 silastic polyethylene pediatric feeding tube with multiple side-holes is inserted 2 cm into the pancreatic duct. The catheter exited via a small enterotomy in the jejunal loop of the distal portion of the hepaticojejunostomy. Totally externalized pancreatic stents were connected to the aspiration bag of a Jackson-Pratt drain to generate negative pressure or to a bile bag for natural drainage.
  Other Names: pancreaticojejunostomy
  Arms: 1
Procedure: natural drainage of pancreatic duct — Natural drainage group
  Other Names: pancreaticojejunostomy
  Arms: 2

SUMMARY:
Pancreaticojejunal anastomosis leakage is a major complication after pancreatoduodenectomy and various technical methods have been examined to improve the situation.However, none of methods have been successful at improving results according to the findings of prospective randomized studies. We propose that active drainage of pancreatic juice using suction drainage might maximize the advantage of a stent and finally reduce pancreaticojejunal anastomosis leakage.

DETAILED DESCRIPTION:
Pancreaticojejunal anastomosis leakage is a major complication after pancreatoduodenectomy and various technical methods have been examined to improve the situation, e.g., pancreatic duct occlusion, anastomosis reinforcement with fibrin glue, placement of an internal stent, and pancreaticogastrostomy. However, none of these methods have been successful at improving results according to the findings of prospective randomized studies. Some retrospective studies have reported a low pancreatic fistula rate when a catheter is inserted into the pancreatic duct to externally drain pancreatic juice. Furthermore, a recent prospective randomized trial showed that external drainage of the pancreatic duct decreased the rate of pancreatic fistula formation indicating that diverting pancreatic juice from an anastomosis can theoretically reduce the incidence of pancreaticojejunostomy anastomotic leakage. We propose that active drainage of pancreatic juice using suction drainage might maximize the advantage of a stent and finally reduce pancreaticojejunal anastomosis leakage.

We will enroll all patients who underwent duct-to-mucosa pancreaticojejunostomy reconstruction after pancreatoduodenectomy, and randomly allocate them to two groups of closed suction drainage group (CD group) and natural drainage group (ND group) just after operations.

Preoperative demographic and clinical data, and surgical procedure, pathologic diagnosis, postoperative course and complications details were collected prospectively.

The primary study endpoints were; pancreatic fistula rates, severity of pancreatic fistulas, postoperative complications, postoperative length of hospital stay, and hospital mortality rate. Pancreatic fistula was defined as any measurable drainage from an operatively placed drain (or a subsequently placed percutaneous drain) on or after postoperative day 3, with an amylase content greater than 3 times the upper limit of normal serum amylase level (i.e., >300 IU/L)(International Study Group for Pancreatic Fistulas (ISGPF) definition) or on or after postoperative week 1 drainage of more than 30 mL of fluid with an amylase level higher than 600 U/dL(Seoul National University Hospital (SNUH) definition). In addition, fistula severity was graded as A, B, C according to ISGPF clinical criteria as follows; grade A fistula - a transient, asymptomatic fistula with only elevated drain amylase levels and treatments or deviation in clinical management are not required; grade B fistula - a symptomatic, clinically apparent fistula requiring diagnostic evaluation and therapeutic management; and grade C fistula - a severe, clinically significant fistula requiring a major deviations in clinical management and unequivocal aggressive therapeutic interventions. Major pancreatic leakage was defined as drainage of more than 200 mL of fluid or the development of an intra-abdominal abscess.

ELIGIBILITY:
Inclusion Criteria:

* All patients who undergo duct-to-mucosa pancreaticojejunostomy reconstruction after pancreatoduodenectomy in our institution

Exclusion criteria:

* less than 15 years old, or older than 85 years old

Ages: 15 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2007-03; Primary Completion 2009-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sun-Whe Kim, MD., PhD., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Background] Hamanaka Y, Suzuki T. Total pancreatic duct drainage for leakproof pancreatojejunostomy. Surgery. 1994 Jan;115(1):22-6. PMID 8284756
- [Background] Mok KT, Wang BW, Liu SI. Management of pancreatic remnant with strategies according to the size of pancreatic duct after pancreaticoduodenectomy. Br J Surg. 1999 Aug;86(8):1018-9. doi: 10.1046/j.1365-2168.1999.01206.x. No abstract available. PMID 10460636
- [Background] Poon RT, Fan ST, Lo CM, Ng KK, Yuen WK, Yeung C, Wong J. External drainage of pancreatic duct with a stent to reduce leakage rate of pancreaticojejunostomy after pancreaticoduodenectomy: a prospective randomized trial. Ann Surg. 2007 Sep;246(3):425-33; discussion 433-5. doi: 10.1097/SLA.0b013e3181492c28. PMID 17717446
- [Background] Lee SE, Yang SH, Jang JY, Kim SW. Pancreatic fistula after pancreaticoduodenectomy: a comparison between the two pancreaticojejunostomy methods for approximating the pancreatic parenchyma to the jejunal seromuscular layer: interrupted vs continuous stitches. World J Gastroenterol. 2007 Oct 28;13(40):5351-6. doi: 10.3748/wjg.v13.i40.5351. PMID 17879405

RESULTS

PARTICIPANT FLOW:
Groups:
- Closed Suction Drainage Group: closed suction drainage group (CD group)
- Natural Drainage Group: natural drainage group (ND group)
Period: Overall Study
Arm/Group | Closed Suction Drainage Group | Natural Drainage Group
Started | 86 | 82
Completed | 86 | 82
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Closed Suction Drainage Group | Natural Drainage Group | Total
Number analyzed (Participants) | 86 | 82 | 168
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 59 | 49 | 108
  >=65 years | 27 | 33 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.7 (10.1) | 61.4 (11.1) | 61.2 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 27 | 64
  Male | 49 | 55 | 104
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 86 | 82 | 168

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Pancreatic Fistula
Description: pancreatic fistula rate is stratified according to ISGPF criteria.
  Grade A; No major impact Grade B; Clinically relevant fistula, specific treatment may be required Grade C; Most severe form of fistula, with a high mortality rate
Time Frame: postoperative 1 week
Measure: Number; unit: participants
Arm/Group | Closed Suction Drainage Group | Natural Drainage Group
Number analyzed (Participants) | 86 | 82
participants | 9 | 8

2. Secondary Outcome: Severity of Pancreatic Fistulas
Time Frame: 2 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Closed Suction Drainage Group | Natural Drainage Group
Serious Adverse Events (participants affected / at risk) | 0/86 | 0/82
Other Adverse Events (participants affected / at risk) | 0/86 | 0/82

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No